CLINICAL TRIAL: NCT04969653
Title: The Incidence of Venous Thromboembolism in Atopic Dermatitis: A Matched Cohort Analysis in UK Primary Care
Brief Title: The Incidence of Venous Thromboembolism in Atopic Dermatitis
Status: Completed | Type: Observational
Sponsor: Momentum Data (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: P046
Record Dates: First submitted 2021-07-01; First posted 2021-07-21 (Actual); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-10

CONDITIONS: Venous Thromboembolism; Atopic Dermatitis; Pulmonary Embolism; Deep Vein Thrombosis; Allergic Rhinitis; Allergy to House Dust Mite; Allergy to Animal Dander; Food Allergy; Cows Milk Allergy
MeSH Terms: conditions — Venous Thromboembolism; Dermatitis, Atopic; Pulmonary Embolism; Venous Thrombosis; Rhinitis, Allergic; Dust Mite Allergy; Food Hypersensitivity; Milk Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: All adults with an episode of active atopic dermatitis at any point between 1st Jan 2010 to 1st Jan 2015 will be included for analysis.
  Interventions: Other: Exposure of venous thromboembolism
- Controls: Adults without atopic dermatitis or other skin conditions matched to cases by age, gender, and duration of practice registration.
  Interventions: Other: Exposure of venous thromboembolism

INTERVENTIONS:
Other: Exposure of venous thromboembolism — Composite of pulmonary embolism and deep vein thrombosis

SUMMARY:
This study aims to investigate the incidence of venous thromboembolism in people who are diagnosed with atopic dermatitis.

DETAILED DESCRIPTION:
The aim of this study is to examine whether venous thromboembolism is higher in people with atopic dermatitis compared and those without and to explore the risk in particular subgroups of people with AD such as those with higher body mass index or using oestrogen containing contraceptives. Such insights will be valuable for clinicians in advising patients with atopic dermatitis regarding venous thromboembolism prevention and detection and when selecting atopic dermatitis treatments.

ELIGIBILITY:
Inclusion Criteria:

* All eligible adult people (aged ≥ 18) registered with GP practices contributing data to OPCRD between January 1, 2010 and January 1, 2020, were eligible for inclusion in the study.

Exclusion Criteria:

* People with less than 5 years potential follow up. People with atopic dermatitis that was not active atopic dermatitis during the study period. People without atopic dermatitis but diagnosed with other skin conditions.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will use routinely collected and collated data from OPCRD to provide a broadly representative sample of the population of the UK.
Sampling Method: Non-Probability Sample
Enrollment: 754745 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew McGovern, MD, Study Director — Momentum Data Ltd
Locations (1):
- Momentum Data Ltd, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
OPCRD data can be accessed by bone fide researchers for specific research projects, subject to approval by Anonymised Data Ethics & Protocol Transparency (ADEPT) Committee. The data utilised for this study cannot be made available without such approval.
Supporting Information: Study Protocol
Time Frame: The data will be available subject to approvals for two years after the study publication date
Access Criteria: Data sharing is subject to ADEPT committee approval

REFERENCES:
- [Result] Warren RB, Basey V, Lynam A, Curtis C, Ardern-Jones MR. The risk of venous thromboembolism in atopic dermatitis: a matched cohort analysis in UK primary care. Br J Dermatol. 2023 Sep 15;189(4):427-436. doi: 10.1093/bjd/ljad212. PMID 37418627

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cases | Controls
Started | 150975 | 603770
Completed | 150975 | 603770
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cases | Controls | Total
Number analyzed (Participants) | 150975 | 603770 | 754745
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 40.0 [23.0 to 62.0] | 41.0 [23.0 to 62.0] | 41.0 [23.0 to 62.0]
Age, Customized [Count of Participants; unit: Participants]
  18-29 | 54634 | 213727 | 268361
  30-39 | 20599 | 80118 | 100717
  40-49 | 17903 | 80211 | 98114
  50-59 | 15765 | 61343 | 77108
  60-69 | 17375 | 71571 | 88946
  70-79 | 15081 | 58452 | 73533
  80+ | 9618 | 38348 | 47966
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89093 | 356311 | 445404
  Male | 61882 | 247459 | 309341
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 87748 | 331717 | 419465
  Asian or Asian British | 12635 | 38388 | 51023
  Black or Black British | 2021 | 7903 | 9924
  Mixed | 1396 | 4281 | 5677
  Not stated | 4638 | 21349 | 25987
  Other | 7503 | 26907 | 34410
  Missing | 35034 | 173225 | 208259
GP visit in last 12 months [Count of Participants; unit: Participants]
  Yes | 146440 | 536511 | 682951
  No | 4535 | 67259 | 71794
BMI [Count of Participants; unit: Participants]
  < 18.5 Underweight | 5931 | 24532 | 30463
  18.5-24.9 Normal weight | 46458 | 174953 | 221411
  25-29.9 Overweight | 43720 | 159607 | 203327
  30-34.9 Class I obesity | 21317 | 77432 | 98749
  35-39.9 Class II obesity | 8711 | 30258 | 38969
  40+ Class III obesity | 5353 | 17515 | 22868
  Missing | 19485 | 119473 | 138958
Smoking status [Count of Participants; unit: Participants]
  Never | 45,152 | 189,107 | 234259
  Current | 27,173 | 116,895 | 144068
  Ex-smoker | 74,860 | 255,950 | 330810
  Passive | 770 | 1,904 | 2674
  Missing | 3020 | 39914 | 42934
Alcohol status [Count of Participants; unit: Participants]
  None | 47083 | 170663 | 217746
  Within limits | 58905 | 226953 | 285858
  Excess | 18660 | 64716 | 83376
  Harmful | 2374 | 8743 | 11117
  Missing | 23953 | 132695 | 156648
Hospital admission [Count of Participants; unit: Participants]
  Yes | 3658 | 11560 | 15218
  No | 147317 | 592210 | 739527

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Diagnosis of Venous Thromboembolism After the Start of Follow-up for Each Person.
Description: To describe the risk of venous thromboembolism (composite of pulmonary embolism and deep vein thrombosis) in people with active AD compared to a matched control population.
Time Frame: 10 years from index date
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 150975 | 603770
Participants | 2576 | 7563

2. Secondary Outcome: Number of Participants With Diagnosis of Pulmonary Embolism After the Start of Follow-up for Each Person
Description: To describe the risk of pulmonary embolism in people with active AD compared to a matched control population.
Time Frame: 10 years from index date
Measure: Count of Participants; unit: Participants
Groups:
- Cases: All adults with an episode of active atopic dermatitis at any point between 1st Jan 2010 to 1st Jan 2015 will be included for analysis.
  Exposure of pulmonary embolism
- Controls: Adults without atopic dermatitis or other skin conditions matched to cases by age, gender, and duration of practice registration.
  Exposure of pulmonary embolism
Arm/Group | Cases | Controls
Number analyzed (Participants) | 150975 | 603770
Participants | 797 | 2942

3. Secondary Outcome: Number of Participants With Diagnosis of Deep-vein Thrombosis After the Start of Follow-up for Each Person
Description: To describe the risk of deep-vein thrombosis in people with active AD compared to a matched control population.
Time Frame: 10 years from index date
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 150975 | 603770
Participants | 1887 | 4934

4. Secondary Outcome: Number of Male Participants With Diagnosis of Risk of Venous Thromboembolism After the Start of Follow-up for Each Person
Description: To explore the risk of VTE stratified by the male sex at the baseline in people with active AD compared to a matched control population.
Time Frame: 10 years from index date
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 61882 | 247459
Participants | 1070 | 3170

5. Secondary Outcome: Number of Female Participants With Diagnosis of Risk of Venous Thromboembolism After the Start of Follow-up for Each Person
Description: To explore the risk of VTE stratified by the female sex at the baseline in people with active AD compared to a matched control population.
Time Frame: 10 years from index date
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 89093 | 356311
Participants | 1506 | 4393

6. Secondary Outcome: Number of Participants Aged 18-44 With Diagnosis of Venous Thromboembolism After the Start of Follow-up for Each Person
Description: To explore the risk of VTE stratified by those aged 18-44 at the baseline in people with active AD compared to a matched control population.
Time Frame: 10 years from index date
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 84253 | 337007
Participants | 503 | 1592

7. Secondary Outcome: Number of Participants Aged 45-64 With Diagnosis of Venous Thromboembolism After the Start of Follow-up for Each Person
Description: To explore the risk of VTE stratified by those aged 45-64 at the baseline in people with active AD compared to a matched control population.
Time Frame: 10 years from index date
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 33497 | 133987
Participants | 639 | 1858

8. Secondary Outcome: Number of Participants Aged ≥65 With Diagnosis of Venous Thromboembolism After the Start of Follow-up for Each Person
Description: To explore the risk of VTE stratified by those aged ≥65 at the baseline in people with active AD compared to a matched control population.
Time Frame: 10 years from index date
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 33225 | 132776
Participants | 1434 | 4113

9. Secondary Outcome: Number of Participants BMI <30 With Diagnosis of Venous Thromboembolism After the Start of Follow-up for Each Person
Description: To explore the risk of VTE stratified by those with a BMI <30 at the baseline with active AD compared to a matched control population.
  Patients with active AD and missing BMI are excluded along with their related matched cases.
  Patients with active AD and no matched controls with BMI recorded are also excluded.
Time Frame: 10 years from index date
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 92915 | 249186
Participants | 1398 | 3188

10. Secondary Outcome: Number of Participants BMI ≥30 With Diagnosis of Venous Thromboembolism After the Start of Follow-up for Each Person
Description: To explore the risk of VTE stratified by those with a BMI ≥30 at the baseline in people with active AD compared to a matched control population.
  Patients with active AD and missing BMI are excluded along with their related matched cases.
  Patients with active AD and no matched controls with BMI recorded are also excluded.
Time Frame: 10 years from index date
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 23725 | 36835
Participants | 685 | 760

11. Secondary Outcome: Number of Female Participants Aged 18-44 Using Oestrogen Contraceptive With Diagnosis of Venous Thromboembolism After the Start of Follow-up for Each Person
Description: To explore the risk of VTE stratified by oestrogen contraceptive use in females aged 18-44 years at the baseline in people with active AD compared to a matched control population.
Time Frame: 10 years from index date
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 4917 | 6925
Participants | 31 | 34

12. Secondary Outcome: Number of Participants Having History of an Allergic Condition With Diagnosis of Venous Thromboembolism After the Start of Follow-up for Each Person
Description: To explore risk of VTE stratified by the presence, or absence of allergic conditions at baseline in people with active AD compared to a matched control population.. Allergic conditions will comprise common allergies; allergic rhinitis, allergy to dust mites or animal dander, and food allergies e.g., nut, fruit, shellfish, eggs and cows' milk allergies. Medication and other allergies will not be included.
Time Frame: 10 years from index date
Measure: Count of Participants; unit: Participants
Arm/Group | Cases | Controls
Number analyzed (Participants) | 18742 | 25088
Participants | 193 | 203

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Cases | Controls
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-05): https://cdn.clinicaltrials.gov/large-docs/53/NCT04969653/Prot_SAP_000.pdf